CLINICAL TRIAL: NCT01121107
Title: Left Atrial Pressure Monitoring to Optimize Heart Failure Therapy Study
Brief Title: Left Atrial Pressure Monitoring to Optimize Heart Failure Therapy
Acronym: LAPTOP-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: G090084
Record Dates: First submitted 2010-05-05; First posted 2010-05-12 (Estimated); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Heart Failure
Keywords: Heart Failure; Decompensated Heart Failure; Acute Decompensated Heart Failure; Hemodynamic Monitoring; Implantable Pressure Monitor; Left Atrial Pressure Monitoring
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Left Atrial Pressure Monitoring System (Experimental): Left Atrial Pressure (LAP) Monitoring System
  Interventions: Device: Left Atrial Pressure Monitoring System; Device: Patient Advisory Module
- Patient Advisor Module (Active Comparator): Patient Advisory Module
  Interventions: Device: Patient Advisory Module

INTERVENTIONS:
Device: Left Atrial Pressure Monitoring System — Left atrial lead is placed for ambulatory monitoring of left atrial pressure
  Arms: Left Atrial Pressure Monitoring System
Device: Patient Advisory Module — Handheld device that provides medication reminders

SUMMARY:
The purpose of this clinical study is to evaluate the safety and clinical effectiveness of use of a physician-directed, patient self-management system, guided by left atrial pressure measurements, for use in patients with heart failure. The system allows patients to adjust their HF medications daily based on a physician-directed prescription plan and their current HF status, similar to the manner in which diabetes patients manage their insulin therapy. The goal of the LAPTOP-HF study is to demonstrate reductions in episodes of worsening heart failure (HF) and hospitalizations in patients who are managed with the left atrial pressure (LAP) management system (treatment group) versus those who receive only the current standard of care (control group).

DETAILED DESCRIPTION:
The Sponsor believes that direct measurements from your heart may provide an accurate, reliable and medically acceptable way of better managing your heart failure prior to your noticing symptoms or being hospitalized. This may enable you and your doctor to take preventative measures, by fine tuning your care including more frequently adjusting your medications with a goal of avoiding hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Have ischemic or non-ischemic cardiomyopathy with either a history of reduced or preserved ejection fraction and heart failure for at least 6 months.
* NYHA Class III documented at screening visit.
* Be receiving appropriate medical therapy for heart failure as per ACC/AHA guidelines (such as diuretic, angiotensin-converting enzyme (ACE) inhibitor or angiotensin receptor blocker (ARB) and beta-blocker) for at least 3 months prior to the randomization visit. Subject has been on stable medications maximized to the subject's tolerance of ACE or ARB and beta-blockers as determined by the study investigator for at least 30 days prior to randomization. Stable is defined as no more than a 100% increase or 50% decrease in dose. These criteria may be waved if a subject is intolerant of ACE, ARB or beta-blockers, or these agents are not indicated under the Guidelines. Such intolerance or lack of indications must be documented.
* Have a minimum of one (1) prior hospital admission within the last 12 months for acute exacerbation of HF of at least one (1) calendar date change duration requiring intravenous or invasive HF therapy. If CRT device previously implanted, the heart failure hospitalization must be ≥ 30 days after CRT implantation. Alternatively, if patients have not had a heart failure hospitalization within the prior 12 months, they must have an elevated Brain Natriuretic Peptide (BNP) level of at least 400pg/ml or an N-terminal pro-BNP (NT-proBNP) level of at least 1,500pg/ml, according to local measurement at the time of screening (within 30 days of the screening visit/consent)
* Provide informed consent for study participation and be willing and able to comply with the required tests, treatment instructions and follow-up visits.
* Are able to schedule Therapy Initiation within two weeks. Enrollment/Randomization may be delayed until this criterion is met.

Exclusion Criteria:

* Are under the age of 18 years.
* Are pregnant.
* Have intractable HF with resting symptoms despite maximal medical therapy (persistent NYHA Class IV and ACC/AHA HF Stage D). This includes patients receiving continuous or intermittent outpatient intravenous vasoactive medications (e.g., IV inotropes, IV vasodilators), patients treated with a ventricular assist device (VAD), and patients who have received a cardiac transplant or are listed for cardiac transplantation and likely to be transplanted within 12 months - even if their functional status has improved to NYHA Class III. Patients listed for cardiac transplantation who are not likely to be transplanted within 12 months and who have improved to NYHA Class III without outpatient IV vasoactive medications or a VAD are eligible for the study, if they meet the other inclusion/exclusion criteria.
* Have a resting systolic blood pressure < 80 or > 180 mmHg.
* Have an acute MI, Acute Coronary Syndrome, Percutaneous Coronary Intervention (PCI), new cardiac rhythm management device (Pacemaker, ICD, and CRT), CRM system revision, lead extraction or cardiac or other major surgery within 40 days.
* Have known coexisting, untreated, hemodynamically severe stenotic valve lesions, vegetations, hypertrophic cardiomyopathy with significant resting or provoked subaortic gradient, acute myocarditis, tamponade, or large pericardial effusion.
* Have an Atrial Septal Defect or Patent Foramen Ovale (with more than trace shunting on color Doppler or intravenous bubble study) or surgical correction of significant congenital heart disease involving atrial septum such as PFO or ASD closure device.
* Have a Stroke or Transient Ischemic Attack within 6 months.
* Have inadequate vascular access for device implantation.
* Have baseline 2-D echocardiographic evidence of, or history of, unresolved left atrial or ventricular thrombus.
* Have a recent (within 6 months) or persistent deep venous thrombosis, pulmonary or systemic thromboembolism.
* Have a life expectancy < 1 year due to another illness.
* Have coagulopathy or uninterruptible anticoagulation therapy or contraindication for all of the forms of antiplatelet/anticoagulant treatments anticipated in the protocol.
* Have an Estimated Glomerular Filtration Rate that remains < 30 ml/min/1.73 M2 by the MDRD method.
* Have a Liver Function Test > 3 times upper limit of normal.
* Have Severe Pulmonary Disease producing frequent hospitalizations for respiratory distress and requiring continuous home oxygen.
* Have pulmonary hypertension with a pulmonary artery systolic pressure of greater than or equal to 80 mm/Hg on screening echocardiogram.
* Have an active infection requiring systemic antibiotics.
* Have a history of active drug addiction, active alcohol abuse, or psychiatric hospital admission for psychosis within the prior 2 years.
* Are currently participating in a clinical investigation that includes an active treatment arm.
* Are unable to demonstrate understanding and capability of using the PAM patient advisory module appropriately.
* Patient does not have access to a telephone line usable for remote PAM follow-up or electrical outlet for recharging PAM.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 486 (Actual)
Dates: Start 2010-04; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Freedom from study-related major adverse cardiovascular and neurological events (MACNE) | 12 months
  Safety will be demonstrated by evaluating the freedom from study-related (procedure or device) major adverse cardiovascular and neurological events (MACNE) in the Treatment group at 12 months from Randomization. The secondary safety endpoint is a non-inferiority analysis of the relative risk (RR) of All-Cause MACNE between the Treatment group and the Control group.
Reduction in Relative Risk of Heart Failure Hospitalization | event driven
  Effectiveness will be determined by evaluating the reduction in the relative risk (RRR) of Heart Failure MACNE between the Treatment and Control groups from randomization. The secondary effectiveness endpoints are days alive and out of the hospital for HF through 12 months after the randomization and all-cause death at 12 months from the randomization.

CONTACTS AND LOCATIONS:
Overall Officials: Leway Chen, M.D., Principal Investigator — University of Rochester, Strong Memorial Hospital, Rochester, NY; Leslie Saxon, M.D., Principal Investigator — USC University Hospital, Los Angeles, CA; John P. McKenzie III, MD, Principal Investigator — Glendale Memorial Hospital and Medical Center, Glendale, CA; Steven Bailin, MD, Principal Investigator — Iowa Heart Center, Des Moines, IA; Dhanunjaya Lakkireddy, MD, Principal Investigator — Mid-America Cardiology Associates, PC, Kansas City, KS; Hamang Patel, MD, Principal Investigator — Ochsner Health System; Ayesha Hasan, MD, Principal Investigator — Ohio State University; Philip B. Adamson, MD, Principal Investigator — Oklahoma Cardiovascular Research Group, Oklahoma City, OK; Steve Hsu, MD, Principal Investigator — Shands Jacksonville, Jacksonville, FL; John Ferguson, MD, Principal Investigator — University of Virginia Medical Center, Charlottesville, VA; Steven Krueger, MD, Principal Investigator — Bryan LGH Heart Institute, Lincoln, NE; Andrew Civitello, MD, Principal Investigator — Texas Heart Institute, Houston, TX; Theo Meyer, MD, Principal Investigator — University of Massachusetts Medical Center, Worcester, MA; Stephen W Halpern, MD, Principal Investigator — Radiant Research, Santa Rosa, CA; Rami Alharethi, MD, Principal Investigator — Intermountain Heart Rhythm Specialists, Murray, UT; Otfried Neidermaier, MD, Principal Investigator — Northeast Ohio Cardiovascular Specialists, Akron, OH; Marlo Leonen, MD, Principal Investigator — Trinity Health-Michigan d/b/a Michigan Heart, Ann Arbor, MI; Peter Pak, MD, Principal Investigator — Pacific Heart Institute, Santa Monica, CA; Maria Rosa Costanzo, MD, Principal Investigator — Advocate Health and Hospitals Corporation, Oakbrook Terrace, IL; Nasir Sulemanjee, MD, Principal Investigator — Aurora Sinai Medical Center, Milwaukee, WI; John Gurley, MD, Principal Investigator — University of Kentucky, Lexington, KY; Barry Cabuay, MD, Principal Investigator — Minneapolis Heart Institute, Minneapolis, MN; Stephen Winters, MD, Principal Investigator — Morristown Memorial Hospital, Morristown, NJ; Wilson Tang, MD, Principal Investigator — The Cleveland Clinic Foundation, Cleveland, OH; Kimberly Parks, MD, Principal Investigator — Massachusetts General Hospital; David Delurgio, MD, Principal Investigator — Emory University Hospital, Atlanta, GA; Niraj Sharma, MD, Principal Investigator — St. Joseph's Hospital, Atlanta, GA; Frank McGrew, MD, Principal Investigator — Baptist Memorial Hospital, Memphis, TN; Thomas O'Brien, MD, Principal Investigator — The Lindner Center, Cincinnati, OH; Peter Fattal, MD, Principal Investigator — MidMichigan Physicians Group, Midland, MI; Aaron Berman, MD, Principal Investigator — Beaumont Hospital, Royal Oak, MI; John Herre, MD, Principal Investigator — Sentara Norfolk General Hospital, Norfolk, VA; James Maher, MD, Principal Investigator — University of Medicine & Dentistry of New Jersey, Newark, NJ; Michael Craig, MD, Principal Investigator — Medical University of South Carolina; Robert Gordon, MD, Principal Investigator — Northwestern Memorial Hospital, Chicago, IL; Daniel J Lenihan, MD, Principal Investigator — Vanderbilt University Hospital, Nashville, TN; Thomas J. Heywood, MD, Principal Investigator — Scripps Green Hospital, La Jolla, CA; Rohit Mehta, MD, Principal Investigator — Sanger Clinic, Charlotte, NC; Daniel Landa, MD, Principal Investigator — St. Jude Hospital, Fullerton, CA; Anju Nohria, MD, Principal Investigator — Brigham and Women's Hospital, Boston, MA; Mark Everley, MD, Principal Investigator — St. Luke's Hospital, Kansas City, MO; Richard Troughton, MD, Principal Investigator — Christchurch Hospital, Christchurch, New Zealand; George Sokos, MD, Principal Investigator — Allegheny Singer Research Institute, Pittsburgh, PA; Paul Coffeen, MD, Principal Investigator — Austin Heart, Austin, TX; Ashish Gupta, MD, Principal Investigator — Cardiovascular Consultants Ltd, Phoenix, AZ; Lawrence Czer, MD, Principal Investigator — Cedars-Sinai Medical Center, Los Angeles, CA; Joseph Rogers, MD, Principal Investigator — Duke University Medical Center, Durham, NC; Tarek Nossuli, MD, Principal Investigator — Lancaster General Hospital, Lancaster, PA; Dusan Kocovic, MD, Principal Investigator — Main Line Health Center/Lankenau Hospital, Wynnewood, PA; John Boehmer, MD, Principal Investigator — Penn State Milton S. Hershey Medical Center, Hershey, PA; Jason Zagrodzky, MD, Principal Investigator — Texas Cardiac Arrhythmia, Austin, TX; Jerry Estep, MD, Principal Investigator — The Methodist Hospital, Houston, TX; Mauricio Hong, MD, Principal Investigator — VA Medical Center Cleveland, Cleveland, OH; Michael Pham, MD, Principal Investigator — VA Palo Alto Medical Center, Palo Alto, CA; Alaa Shalaby, MD, Principal Investigator — VA Pittsburgh Healthcare System, Pittsburgh, PA; Zi-Juan Xu, MD, Principal Investigator — Sutter Memorial Hospital, Sacramento, CA; Liviu Klein, MD, Principal Investigator — University of California at San Francisco; Jerry John, MD, Principal Investigator — McKay-Dee Heart Services, Ogden, UT; Pranav Loyalka, MD, Principal Investigator — Memorial Hermann Hospital, Houston, TX; Greg Ewald, MD, Principal Investigator — Washington University School of Medicine; Debbie A. Rinde-Hoffman, MD, Principal Investigator — Tampa General Hospital, Tampa, FL; Frank Smart, MD, Principal Investigator — Louisiana State University Health Sciences Center, New Orleans, LA; Kelly McCants, MD, Principal Investigator — Jewish Hospital, Louisville, KY; Jacob Abraham, MD, Principal Investigator — Providence Heart and Vascular Institute, Portland, OR
Locations (64):
- United States (63):
  - Cardiovascular Consultants Ltd, Phoenix, Arizona
  - St. Jude Hospital, Fullerton, California
  - Glendale Memorial Hospital and Medical Center, Glendale, California
  - Scripps Green Hospital, La Jolla, California
  - USC University Hospital, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - VA Palo Alto Medical Center, Palo Alto, California
  - Sutter Memorial Hospital, Sacramento, California
  - University of California at San Francisco, San Francisco, California
  - Pacific Heart Institute, Santa Monica, California
  - Radiant Research, Santa Rosa, California
  - Shands Jacksonville, Jacksonville, Florida
  - Tampa General Hospital, Tampa, Florida
  - The Emory Clinic - Crawford Long Hospital, Atlanta, Georgia
  - St. Joseph's Hospital, Atlanta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Advocate Health and Hospitals Corporation, Oakbrook Terrace, Illinois
  - Iowa Heart Center, Des Moines, Iowa
  - Mid-America Cardiology Associates, PC, Kansas City, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Louisiana State University Health Sciences Center, New Orleans, Louisiana
  - Ochsner Medical Center, New Orleans, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Massachusettts Medical Center, Worcester, Massachusetts
  - Trinity Health - Michigan d/b/a Michigan Heart, Ann Arbor, Michigan
  - MidMichigan Physicians Group, Midland, Michigan
  - Beaumont Hospital, Royal Oak, Royal Oak, Michigan
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - St. Luke's Hospital, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Bryan LGH Heart Institute, Lincoln, Nebraska
  - Morristown Memorial Hospital, Morristown, New Jersey
  - University of Medicine & Dentistry of New Jersey, Newark, New Jersey
  - University of Rochester, Rochester, New York
  - Sanger Clinic, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Northeast Ohio Cardiovascular, Akron, Ohio
  - The Linder Center, Cincinnati, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - VA Medical Center Cleveland, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Oklahoma Cardiovascular Research Group, Oklahoma City, Oklahoma
  - Providence Heart and Vascular Institute, Portland, Oregon
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Lancaster Heart Foundation, Lancaster, Pennsylvania
  - Allegheny Singer Research Institute, Pittsburgh, Pennsylvania
  - VA Pittsburgh Healthcare System, Pittsburgh, Pennsylvania
  - Main Line Health Heart Center: Lankenau Hospitals, Wynnewood, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Baptist Memorial Hospital, Memphis, Tennessee
  - Vanderbilt Medical Center, Nashville, Tennessee
  - Austin Heart, Austin, Texas
  - Texas Cardiac Arrhythmia Research Foundation, Austin, Texas
  - Memorial Hermann Hospital, Houston, Texas
  - Methodist Hospital Research Institute, Houston, Texas
  - Texas Heart Institute, Houston, Texas
  - Intermountain Heart Rhythm Specialists, Murray, Utah
  - McKay-Dee Heart Services, Ogden, Utah
  - University of Virginia Medical Center, Charlottesville, Virginia
  - Sentara Hospitals and Sentara Cardiovascular Research Institute, Norfolk, Virginia
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
- Christchurch Hospital, Christchurch, New Zealand